CLINICAL TRIAL: NCT01988220
Title: The Effects of Lower Extremity Sensory Retraining Treatment in Individuals With Post-stroke Sensory Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yocheved Laufer (Other)
Collaborators: Clalit Health Services, Haifa and West Galilee (Other)
Responsible Party: Sponsor-Investigator, Yocheved Laufer, Chair, Physical Therapy Department, University of Haifa
Organization: University of Haifa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHai012013
Record Dates: First submitted 2013-11-05; First posted 2013-11-20 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Stroke; Sensory Deficits
Keywords: stroke; sensory deficit; sensory retraining; perceptual learning; lower extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sensory retraining (Experimental): sensory identification and discrimination training. using different attention and sensation modalities for sensory retraining
  Interventions: Other: sensory retraining
- repeated exposure to sensory input (Active Comparator)
  Interventions: Other: repeated sensory input

INTERVENTIONS:
Other: sensory retraining
  Other Names: perceptual learning; sensory reeducation
  Arms: sensory retraining
Other: repeated sensory input — sensory stimulation without attentive learning focus
  Arms: repeated exposure to sensory input

SUMMARY:
Background: It is estimated that 50%-85% of individuals post stroke demonstrate sensory deficits. Sensory impairments are often overlooked in the therapeutic setting, although they lead to slower motor recovery.

Working hypothesis: The overall goal of this study is to examine the effectiveness of a sensory discrimination reeducation oriented therapeutic program to the lower limb of stroke patients with sensory impairments. We assume that subjects to both groups will make progress, which will be more significant in the experimental group.

Methods: Study population and design: Sixty individuals with chronic sensory impairment following a stroke will be recruited. Patients will be randomly assigned to sensory retraining treatment or to sensory stimulation treatment. Treatment will consist of ten 45 minute long intervention sessions, carried out within a 6 weeks period, and a home exercise program. The person conducting the assessments will be blind to the treatment allocation of the subjects. Outcome measures: The efficacy of the intervention will be determined in relation to the International Classification of Functionality (ICF) developed by the World Health Organization and will include assessments at the three domains defined by this model: 1. Body structure and function - determined by measures of the sensory capacity of the lower more affected limb; 2. Activities - determined by measures of balance and gait; 3. Participation - determined by measures of well-being and social reintegration.

Two new outcome measures, for ankle and knee position sense and for texture discrimination of the foot, will be developed within this study. Data reliability measures on healthy population, and test - retest measures in post stroke population with be collected.

Intervention: The experimental group will be treated by a perception learning oriented protocol for sensory reeducation, to improve identification, localization and discrimination of sensory stimuli, including electrical stimulation, texture and hardness discrimination and position sense training. The control group will receive the same stimuli without the attentive learning and discriminating component.

Importance: Scientific proof and focused recommendations for a potent therapeutic method for the post-stroke population, allowing them better participation and quality of life.

Key words: Stroke, sensory impairment, perceptual learning, lower limb, clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* post stroke
* at least 6 months after stroke
* with sensory deficits in study's screening tests

Exclusion Criteria:

* other neurologic condition
* peripheral neuropathy
* pacemaker
* hemispatial neglect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-12; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Timed Up and Go test | pre - up to a week before intervention, post - after 6 weeks, follow-up - 3 months after
  Standing up from a chair, walking three meters, turning around and coming back to sitting. time is assessed.

SECONDARY OUTCOMES:
Von Frey monofilaments foot identification threshold | screening - one week before pretest, pre - up to one week before intervention, post - 6 weeks after, follow-up - 3 months after
  Assessment of threshold for Von Frey monofilaments identification, using the levels method. Starting with monofilament 5.07, two points will be assessed - dorsal mid foot and anterior mid ankle.

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Alperin, MD, Principal Investigator — Clalit Health Services; Hadas Ofek, PhD student, Study Director — University of Haifa; Yocheved Laufer, Professor, Study Chair — University of Haifa; Uzi Milman, MD, Study Chair — Clalit Health Services
Locations (1):
- Physical therapy clinics Clalit Health services, Haifa District, Israel

REFERENCES:
- [Derived] Ofek H, Alperin M, Knoll T, Livne D, Laufer Y. Explicit versus implicit lower extremity sensory retraining for post-stroke chronic sensory deficits: a randomized controlled trial. Disabil Rehabil. 2023 Jun;45(12):1962-1968. doi: 10.1080/09638288.2022.2080288. Epub 2022 Jun 1. PMID 35649684